CLINICAL TRIAL: NCT01463020
Title: Behavioural Activation-Based Guided Self-Help Treatment Administered Through a Smartphone Application
Brief Title: Behavioural Activation-Based Treatment Administered Through Smartphone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-PC-KHL
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Depression; Smartphone; Behavioural activation; Mindfulness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone delivered BA (Experimental)
  Interventions: Behavioral: Smartphone delivered BA
- Smartphone delivered mindfulness (Active Comparator)
  Interventions: Other: Smartphone delivered mindfulness

INTERVENTIONS:
Behavioral: Smartphone delivered BA — A 8 week behavioural activation therapy delivered through smartphone
  Arms: Smartphone delivered BA
Other: Smartphone delivered mindfulness — A 8 week mindfulness intervention delivered through smartphone
  Arms: Smartphone delivered mindfulness

SUMMARY:
The objective is to test the effects of a smartphone-delivered behavioural activation treatment. Also, a moderator analysis of low and high severity of depressive symptoms will be made. We expect the behavioural activation intervention to be superior to the mindfulness intervention for the participants suffering from high severity of depressive symptoms - and the mindfulness intervention to be better or at least as good as the behavioural activation intervention for the participants suffering from low severity of depressive symptoms.

DETAILED DESCRIPTION:
Major depression is expected to be the disorder with the highest disease burden in high-income countries by the year 2030. The efficacy of behavioural activation in the treatment of major depressive disorders has been established in a number of studies over the last four decades. Furthermore, behavioural activation is an intervention that can largely benefit from the use of new mobile technologies (e.g. smartphones). One important feature of mobile technology is the possibility for the therapist to reach the patient between sessions and thus create direct incentives for behavioural activation in everyday life. Therefore, developing smartphone-based behavioural activation interventions might be a way to develop a cost-effective treatment for people suffering from major depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* depressive symptoms according to DSM-IV
* have access to the Internet and a smartphone
* have good knowledge of the Swedish language

Exclusion Criteria:

* recent (during last 6 weeks) change in psychiatric medication
* presently in any other psychological treatment
* severe depression
* suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Beck Depression Inventory (BDI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.

SECONDARY OUTCOMES:
Quality of Life Inventory (QOLI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Acceptance & Action Questionnaire (AAQ)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Beck Anxiety Inventory (BAI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P)- Change from baseline | Two weeks pre treatment and at six months post treatment.
  Change from baseline in health cost burden and at six months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Study Director — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Ly KH, Truschel A, Jarl L, Magnusson S, Windahl T, Johansson R, Carlbring P, Andersson G. Behavioural activation versus mindfulness-based guided self-help treatment administered through a smartphone application: a randomised controlled trial. BMJ Open. 2014 Jan 9;4(1):e003440. doi: 10.1136/bmjopen-2013-003440. PMID 24413342
- [Derived] Ly KH, Carlbring P, Andersson G. Behavioral activation-based guided self-help treatment administered through a smartphone application: study protocol for a randomized controlled trial. Trials. 2012 May 18;13:62. doi: 10.1186/1745-6215-13-62. PMID 22607302